CLINICAL TRIAL: NCT00495573
Title: Half-life and Pattern of Resolution of Herpes Simplex Virus Type 2 (HSV-2) Shedding After Beginning Acyclovir Treatment
Brief Title: HSV-2 Shedding Resolution After Acyclovir Treatment
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Anna Wald, Principal Investigator, University of Washington
Other Study IDs: 26224-A; P01AI030731 (NIH); R01AI050132 (NIH)
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Acyclovir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, genital swab specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: HSV-2 seropositive subjects who will receive a 5-day course of acyclovir for treatment of a genital herpes recurrence.
  Interventions: Drug: acyclovir
- 2: HSV-2 seropositive subjects who will be observed during a genital herpes recurrence but not receive acyclovir.

INTERVENTIONS:
Drug: acyclovir — 400 mg acyclovir, orally three times a day for 5 days
  Groups: 1

SUMMARY:
The purpose of the study is to evaluate the pattern of viral shedding after beginning treatment with acyclovir for a clinical recurrence of genital herpes and to compare it with the pattern of viral shedding during an untreated clinical recurrence of genital herpes.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the pattern of viral shedding after beginning treatment with acyclovir for a clinical recurrence of genital herpes and to compare it with the pattern of viral shedding during an untreated clinical recurrence of genital herpes.

Participants are asked to visit the University of Washington Virology Research Clinic for an initial screening appointment in which the clinician will ensure eligibility and informed consent will be obtained.

Participants who experience an outbreak during the next year will be asked to call the clinic at the beginning of their next outbreak. The clinician will arrange to admit the participant to the UW General Clinical Research Center (GCRC) for a 5-day hospitalization stay. During hospitalization, participants will take acyclovir (400mg 3 times daily) and genital swabs will be collected every 2 hours during the day and every 4 hours at night for 5 days. After the last swab has been taken, the study nurse at the GCRC will do a final genital exam and the participant will be discharged. Some participants will also be asked to enroll in a control arm during which the same procedures will be followed except they will not take acyclovir during the recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of clinically-evident genital herpes
* 3 or more clinical genital herpes recurrences within the prior 12 months
* HSV-2 seropositive by HSV Western Blot
* Willing and able to comply with study protocol

Exclusion Criteria:

* Pregnancy
* Taking daily antiviral therapy for genital herpes
* HIV seropositive or known immunocompromising medical condition
* Plan to move from the Seattle area within the next year
* Hypersensitivity to or intolerance of acyclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HSV-2 seropositive men and women with a history of at least 3 clinical recurrences of genital herpes within the year prior to the screening visit. Participants will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To calculate the half-life of detectable HSV-2 DNA in genital mucosa during a clinical recurrence of genital herpes, after treatment with acyclovir has begun. | 5 days

SECONDARY OUTCOMES:
To describe the time course, diurnal variation, and pattern of resolution of HSV-2 shedding during both acyclovir-treated and untreated clinical recurrences of genital herpes. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States